CLINICAL TRIAL: NCT05187754
Title: The Effects of Mindfulness-based Breathing Therapy on Perceived Stress, Caregiver Burden and Burnout in Caregivers of Palliative Care Patients: Single-blind, Randomised Controlled Study.
Brief Title: The Effects of Mindfulness-based Breathing Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Assistant Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Caregiver mindfulnes
Record Dates: First submitted 2021-12-13; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Palliative Supportive Care; Care Giving Burden
Keywords: Care Giving Burden; Palliative Supportive Care; Burnout
MeSH Terms: conditions — Caregiver Burden; Burnout, Psychological

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Mindfulness-based breathing therapy program
- Control Group (No Intervention)

INTERVENTIONS:
Other: Mindfulness-based breathing therapy program — Participant caregivers of palliative patients were randomized into the intervention and the control groups. Prior to randomization, participants and nurses were informed online abut the aim of the research and their written consent was obtained. Once the study ended, mindfulness-based breathing therapy were recommended to the patients in the control group. Data were collected online via Google forms survey and the interviews were conducted online via Zoom.
  Arms: Intervention Group

SUMMARY:
Aims and objectives: The aim of this study was to assess the effects of mindfulness-based breathing therapy on the levels of perceived stress, caregiver burden and burnout in caregivers of palliative care patients.

Background: It is extremely important to develop evidence-based strategies to protect the psychological health of caregivers, who are part of palliative care, to increase their quality of life and to facilitate their adaptation to the palliative care process.

Design: This was a prospective, single-blind, randomised controlled study. The study complied with the guidelines of Consolidated Standards of Reporting Trials (CONSORT).

Methods: A total of 100 caregivers were randomly assigned to intervention group (n = 50) and control group (n = 50). This single-blinded randomized controlled trial was conducted at the palliative care unit of a private hospital, between May-November 2021. Personal information form, caregiver strain index (CSI), Zarit burden interview (ZBI) and Maslach Burnout Inventory (MBI) were used for data collection.

DETAILED DESCRIPTION:
3.4. Procedures Participant caregivers of palliative patients were randomized into the intervention and the control groups. Prior to randomization, participants and nurses were informed online abut the aim of the research and their written consent was obtained. Once the study ended, mindfulness-based breathing therapy were recommended to the patients in the control group. Data were collected online via Google forms survey and the interviews were conducted online via Zoom. The Principal Investigator, study statisticians, and study staff, who took part in collecting outcome assessments, were blinded to intervention condition. All the measurement scores were obtained by another researcher nurse blinded to arm allocation.

3.4.1. Control Group Participants in the control group were asked to complete the personal information form, CSI, ZBI and MBI online, and sit in a relaxed position in a quiet environment for 30 minutes for three consecutive days. They completed the CSI, ZBI and MBI as posttest at the end of the third day.

3.4.2. Intervention Group 50 participants in the intervention group were divided into ten groups with five participants in each group. After completing the personal information form online, a meeting time was set for each of the ten groups. Participants were asked to be in a quite environment during the meeting and complete the CSI, ZBI and MBI as pretest via Google forms survey. Each group received mindfulness-based breathing therapy for 30 minutes in three consecutive sessions from an expert on the therapy. At the end of the third session, participants completed the CSI, ZBI and MBI as posttest.

Mindfulness-based breathing therapy sessions started by informing the participants about the content of each session and the relaxation effects of breathing on mind and body to cope with stress. Before the breathing exercise, participants were asked to sit in a relaxed position, loosen buttons and belts, take out shoes and close their eyes. They were suggested to put self-judgment aside, focus on the present moment, their breath and finally on each part of their body. To develop concentration and mental flexibility about their bodies, participants were asked to focus on their bodies in a comprehensive and transient way. They were asked to focus on each part of their body stage by stage, combine their consciousness about their breath and body and feel the breath at each part of their body. During the breathing exercises, participants were asked to focus on, feel and realize their emotions. 'TV screen metaphor' was used to put a distance to their opinions and thoughts. They were asked to think about a situation, which made them anxious and stressful, reflect their experience onto a TV screen and think as if they were watching their experience on TV. A piano song was played as background music during the sessions. After taking deep breath for three times, participants were asked to open their eyes.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary caregivers of palliative patients,
* who were 18 years of age and above,
* Did not have any visual or auditory disabilities, were included to the study

Exclusion Criteria:

* Diagnosed with a known psychiatric illness (delirium, anxiety, panic attack, depression)
* Take another psychological relaxation course or training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Baseline
  The form was developed by the researchers in line with the literature and included questions on sociodemographic characteristics of the participants, such as age, gender and education level
Caregiver Strain Index | Baseline
  CSI was developed by Robinson (1983) to measure the burden of care on caregivers and was adapted to Turkish by Uğur & Fadıloğlu (2010). The scale had 13 items, which were scored on a two-point Likert scale, ranging from yes (1 point) to no (0 point).
Caregiver Strain Index | on the seventh day
  CSI was developed by Robinson (1983) to measure the burden of care on caregivers and was adapted to Turkish by Uğur & Fadıloğlu (2010). The scale had 13 items, which were scored on a two-point Likert scale, ranging from yes (1 point) to no (0 point).
Zarit Burden Interview | baseline
  The scale was developed by Zarit et al (1980) and was adapted to Turkish by İnci and Erdem (2008). The scale included 22 items about the impact of caregiving on the life of caregiver, including the psychological and health status and the social life of the caregiver, economic burden on caregiver and the patient/caregiver relationship. Items were scored on a five-point Likert scale, ranging from 0 (never) to 4 (always)
Zarit Burden Interview | on the seventh day
  The scale was developed by Zarit et al (1980) and was adapted to Turkish by İnci and Erdem (2008). The scale included 22 items about the impact of caregiving on the life of caregiver, including the psychological and health status and the social life of the caregiver, economic burden on caregiver and the patient/caregiver relationship. Items were scored on a five-point Likert scale, ranging from 0 (never) to 4 (always)
Maslach Burnout Inventory (MBI) | baseline
  The Scale was developed by Maslach and Jackson (1981) and was adapted to Turkish by Çapri (2006). The scale was composed of 22 items in three subscales, including emotional exhaustion (items 1, 2, 3, 6, 8, 13, 16 and 20), depersonalization (items 5, 10, 11, 15 and 22) and personal accomplishment (items 4, 7, 9, 12, 17, 18, 19 and 21). Emotional exhaustion and depersonalization subscales had items with negative statements whereas the items in the personal accomplishment subscale were positive
Maslach Burnout Inventory (MBI) | on the seventh day
  The Scale was developed by Maslach and Jackson (1981) and was adapted to Turkish by Çapri (2006). The scale was composed of 22 items in three subscales, including emotional exhaustion (items 1, 2, 3, 6, 8, 13, 16 and 20), depersonalization (items 5, 10, 11, 15 and 22) and personal accomplishment (items 4, 7, 9, 12, 17, 18, 19 and 21). Emotional exhaustion and depersonalization subscales had items with negative statements whereas the items in the personal accomplishment subscale were positive

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No